CLINICAL TRIAL: NCT02277782
Title: Intrathecal Hydromorphone for Labor Analgesia
Acronym: LITH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study drug shortage, COVID related suspension of recruitment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dominique Arce, Instructor of Anaesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014P002384
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
Keywords: Labor; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Hydromorphone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Hydromorphone (Active Comparator): 1.7 mg bupivacaine + 17 mcg fentanyl + 0.05 ml of 0.9% normal saline.
  Interventions: Drug: Hyperbaric bupivacaine; Drug: Fentanyl
- Hydromorphone (Experimental): 1.7 mg bupivacaine + 17 mcg fentanyl + 50 mcg preservative-free hydromorphone (0.05 ml)
  Interventions: Drug: Hydromorphone; Drug: Hyperbaric bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Hydromorphone
  Other Names: Dilaudid
  Arms: Hydromorphone
Drug: Hyperbaric bupivacaine
Drug: Fentanyl

SUMMARY:
The objective of this study is to evaluate the effect of intrathecal hydromorphone on the duration of labor analgesia and the incidence of epidural-associated temperature increase in laboring parturients. We hypothesize that intrathecal administration of longer-acting hydromorphone will:

1. Prolong the duration and improve the quality of analgesia in labor, and
2. Decrease the incidence of epidural-associated temperature increase in labor.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for enrollment if they are healthy, pregnant females between the ages of 18 and 45 years, primiparous, and at term gestation (≥ 37 weeks).

Exclusion Criteria:

* Patients with a Category II or III fetal heart rate tracing, a fetus with intrauterine growth restriction, prolonged rupture of membranes, recent diagnosis of infection of any cause, or in whom dural puncture is contraindicated will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on maternal temperature during labor | 2 years
  The primary outcome measure will be the incidence of maternal temperature increase, defined as an increase in maternal temperature by 1 degree celsius over the baseline temperature recorded prior to the onset of epidural analgesia.

SECONDARY OUTCOMES:
Effect on efficacy of labor analgesia | 2 years
  The secondary outcome measure will be the duration of intrathecal analgesia. Additional outcome measures include the quality of analgesia as recorded by the Visual Analogue Scale score and the need for additional top-ups within 90 min of epidural placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States